CLINICAL TRIAL: NCT06059391
Title: Placebo-Controlled and Randomized Phase 2 Trial of CMV-MVA Triplex Vaccination in HLA-Matched Related Stem Cell Donors to Enhance CMV-Specific Immunity and Prevent CMV Viremia in Recipients After Hematopoietic Stem Cell Transplant
Brief Title: CMV-MVA Triplex Vaccination in HLA-Matched Related Stem Cell Donors for the Prevention of CMV Infection in Patients Undergoing Hematopoietic Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23008; NCI-2023-06837 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23008 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01CA266783 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia; Chronic Myeloid Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid System Neoplasm; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myelofibrosis; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Myelodysplastic Syndromes; Primary Myelofibrosis; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin | interventions — Stem Cell Transplantation; Specimen Handling; Granulocyte Colony-Stimulating Factor; Blood Component Removal; Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is observer-blinded because of the handling of the vaccine and the placebo may vary. The investigators, treating clinicians, participants, and other study staff, including the nurses involved in soliciting or recording of adverse events, will be blinded through the day 180 visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Triplex vaccination) (Experimental): DONORS: Donors receive Triplex vaccine IM on day 0 and then undergo stem cell mobilization with G-CSF on days 5 to 9 and apheresis for peripheral blood stem cell collection on days 10 to 14 per standard of care. Donors may optionally undergo blood sample collection on study.
  RECIPIENTS: Recipients undergo pre-transplant conditioning on days -60 to 0 and undergo HCT with the donor peripheral blood stem cells within 9 weeks of donor vaccination on day 0. Recipients undergo blood sample collection on study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Drug: Granulocyte Colony-Stimulating Factor; Drug: Hematopoietic Cell Transplantation Conditioning Regimen; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Pheresis; Drug: Stem Cell Mobilization Therapy
- Arm II (Placebo) (Placebo Comparator): DONORS: Donors receive placebo IM on day 0 and undergo stem cell mobilization with G-CSF on days 5 to 9 and apheresis for peripheral blood stem cell collection on days 10 to 14 per standard of care. Donors may optionally undergo blood sample collection on study.
  RECIPIENTS: Recipients undergo pre-transplant conditioning on days -60 to 0 and undergo HCT with the donor peripheral blood stem cells within 9 weeks of donor vaccination on day 0. Recipients undergo blood sample collection on study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Drug: Granulocyte Colony-Stimulating Factor; Drug: Hematopoietic Cell Transplantation Conditioning Regimen; Procedure: Pheresis; Drug: Placebo Administration; Drug: Stem Cell Mobilization Therapy

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HCT with donor peripheral blood stem cells
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Granulocyte Colony-Stimulating Factor — Undergo stem cell mobilization with G-CSF
  Other Names: Colony Stimulating Factor 3; Colony-Stimulating Factor (Granulocyte); Colony-Stimulating Factor 3; CSF3; G CSF; G-CSF; GCSF; Granulocyte Colony Stimulating Factor; Pluripoietin
Drug: Hematopoietic Cell Transplantation Conditioning Regimen — Receive pre transplant conditioning
  Other Names: HCT Conditioning Regimen; HSCT Conditioning Regimen; Stem Cell Transplant Conditioning
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
  Other Names: CMV-MVA Triplex Vaccine; Multi-antigen CMV-Modified Vaccinia Ankara Vaccine
  Arms: Arm I (Triplex vaccination)
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Drug: Placebo Administration — Given IM
  Arms: Arm II (Placebo)
Drug: Stem Cell Mobilization Therapy — Undergo stem cell mobilization with G-CSF
  Other Names: Chemomobilization; Hematopoietic Stem Cell Mobilization; Mobilization Therapy; Stem-cell mobilization

SUMMARY:
This phase II clinical trial tests how well the cytomegalovirus-modified vaccinica Ankara (CMV-MVA) Triplex vaccine given to human leukocyte antigens (HLA) matched related stem cell donors works to prevent cytomegalovirus (CMV) infection in patients undergoing hematopoietic stem cell transplant. The CMV-MVA Triplex vaccine works by causing an immune response in the donors body to the CMV virus, creating immunity to it. The donor then passes that immunity on to the patient upon receiving the stem cell transplant. Giving the CMV-MVA triplex vaccine to donors may help prevent CMV infection of patients undergoing stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether multi-peptide CMV-modified vaccinia Ankara vaccine (Triplex) is safe and effective in protecting against CMV events defined as viremia requiring antiviral preemptive therapy (PET) or CMV end organ disease.

SECONDARY OBJECTIVE:

I. To examine if Triplex vaccination of hematopoietic stem cell transplant (HCT) donors has an impact on CMV events.

OUTLINE: Donors are randomized to 1 of 2 arms.

ARM I:

DONORS: Donors receive Triplex vaccine intramuscularly (IM) on day 0 and then undergo stem cell mobilization with granulocyte colony-stimulating factor (G-CSF) on days 5 to 9 and apheresis for peripheral blood stem cell collection on days 10 to 14 per standard of care. Donors may optionally undergo blood sample collection on study.

RECIPIENTS: Recipients undergo pre-transplant conditioning on days -60 to 0 and undergo HCT with the donor peripheral blood stem cells within 9 weeks of donor vaccination on day 0. Recipients undergo blood sample collection on study.

ARM II:

DONORS: Donors receive placebo IM on day 0 and undergo stem cell mobilization with G-CSF on days 5 to 9 and apheresis for peripheral blood stem cell collection on days 10 to 14 per standard of care. Donors may optionally undergo blood sample collection on study.

RECIPIENTS: Recipients undergo pre-transplant conditioning on days -60 to 0 and undergo HCT with the donor peripheral blood stem cells within 9 weeks of donor vaccination on day 0. Recipients undergo blood sample collection on study.

After completion of study treatment, donors follow up on days 90, 180 and 365 after vaccination and recipients follow up on days 14, 28, 42, 56, 70, 100, 140, 180, 270, and 365 after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* DONORS: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* DONORS: Age: 18 and above
* RECIPIENTS: Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* RECIPIENTS: Participant must be willing to comply with study and/or follow-up procedures, including willingness to be followed for one year post-HCT
* RECIPIENTS: Age: 18 and above
* RECIPIENTS: Karnofsky performance score ≥ 70 or ECOG ≤ 2
* RECIPIENTS: Planned HCT for the treatment of the following hematologic malignancies: lymphoma (Hodgkin and Non-Hodgkin), myelodysplastic syndrome, acute lymphoblastic leukemia in first or second remission, acute myeloid leukemia in first or second remission, chronic myelogenous leukemia (in first chronic or accelerated phase, or in second chronic phase), chronic lymphocytic leukemia, myeloproliferative disorders and myelofibrosis. Patients with multiple myeloma are excluded
* RECIPIENTS: CMV seropositive
* RECIPIENTS: Planned related HCT with 8/8 (A, B, C, DRB1) high resolution human leukocyte antigen (HLA) donor allele matching
* RECIPIENTS: Conditioning and immunosuppressive regimens according to institutional guidelines are permitted. Patients may receive myeloablative, reduced intensity, or nonmyeloablative conditioning
* RECIPIENTS: Total bilirubin ≤ 2 X upper limit of normal (ULN) (unless has Gilbert's disease)
* RECIPIENTS: Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* RECIPIENTS: Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* RECIPIENTS: Creatinine clearance of ≥ 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* RECIPIENTS: Left ventricular ejection fraction (LVEF) ≥ 50% Note: To be performed within 45 days prior to day 1 of protocol therapy
* RECIPIENTS: If able to perform pulmonary function tests: forced vital capacity (FVC) and diffusion capacity of carbon monoxide (DLCO) (diffusion capacity) ≥ 50% of predicted (corrected for hemoglobin). If unable to perform pulmonary function tests: oxygen (O2) saturation > 92% on room air Note: To be performed within 45 days prior to day 1 of protocol therapy
* RECIPIENTS: Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV)*, active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR])

  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* RECIPIENTS: Meets other institutional and federal requirements for infectious disease titer requirements Note: Infectious disease testing to be performed within 45 days prior to day 1 of protocol therapy
* RECIPIENTS: Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* RECIPIENTS: Agreement by females and males of childbearing potential* to use an effective method of birth control (hormonal or barrier method) or abstain from heterosexual activity prior to study entry and for up to 90 days post-HCT.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* DONORS: Any prior transplant to day 1 of protocol therapy
* DONORS: Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy
* DONORS: Receipt of any vaccine (licensed or investigational) within 30 days prior to and after of the study vaccine
* DONORS: Unfit to undergo standard stem cell mobilization and apheresis e.g. abnormal blood counts, history of stroke, uncontrolled hypertension
* DONORS: Sickling hemoglobinopathy including hemoglobin S (HbSS), sickle cell trait (HbAS), hemoglobin sickle C disease (HbSC)
* DONORS: Donors with impaired cardiac function are excluded. Electrocardiography is routine for potential HCT donors over 60 years old and those with a history of heart disease. Subjects in whom cardiac function is abnormal (excluding 1st degree branch block, sinus bradycardia, sinus tachycardia or non-specific T wave changes) are ineligible for Triplex vaccination
* DONORS: Positive for HIV, active hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II)
* DONORS: Severe psychiatric illness. Mental deficiency sufficiently severe as to make compliance with the donation procedure unlikely, and making informed consent impossible
* DONORS: Females only: Pregnant or breastfeeding
* DONORS: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* DONORS: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* RECIPIENTS: Any prior investigational CMV vaccine
* RECIPIENTS: Experimental anti-CMV chemotherapy in the last 6 months
* RECIPIENTS: Prior allogeneic (allo) transplant for any condition
* RECIPIENTS: Live attenuated vaccines
* RECIPIENTS: Medically indicated subunit (Engerix-B for HBV; Gardasil for HPV) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
* RECIPIENTS: Allergy treatment with antigens injections
* RECIPIENTS: Alemtuzumab or any equivalent in vivo T-cell depleting agent
* RECIPIENTS: Antiviral medications with known therapeutic effects on CMV such as valganciclovir/ganciclovir (GCV/VAL), foscarnet (FOS), cidofovir, brincidofovir (CMX-001), maribavir. Acyclovir has no known therapeutic efficacy against CMV and is allowable as standard of care to prevent herpes simplex virus (HSV)
* RECIPIENTS: Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment
* RECIPIENTS: Other investigational product - concurrent enrollment in other clinical trials using any investigational new drug (IND) drugs with unknown effects on CMV or with unknown toxicity profiles is prohibited
* RECIPIENTS: Other medications that might interfere with the evaluation of the investigational product
* RECIPIENTS: Diagnosis with autoimmune disease
* RECIPIENTS: Females only: Pregnant women and women who are lactating. The risks of Triplex to pregnant women are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother. Breastfeeding should be discontinued if the mother is enrolled on this study
* RECIPIENTS: Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* RECIPIENTS: Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Time from transplantation to cytomegalovirus (CMV) disease or pre-emptive treatment following CMV reactivation (efficacy) | From hematopoietic stem cell transplantation (HCT) to day 180
  A stratified Cox regression analysis of time to CMV disease or positron emission tomography (PET) following CMV reactivation prior to Day 180 post-HCT will be performed. The estimated hazard ratio and its 95% confidence interval will be calculated. Secondary analyses will include the Fine-Gray model for competing risk.
Occurrence of non-relapse mortality (safety in HCT-recipients) | Up to day 100 post HCT
  A stratified Cox regression analysis of time to CMV disease or PET following CMV reactivation prior to Day 180 post-HCT will be performed. The estimated hazard ratio and its 95% confidence interval will be calculated. Secondary analyses will include the Fine-Gray model for competing risk.
Incidence of severe acute graft versus host disease (aGHVD) (safety in HCT-recipients) | Up to 100 days post HCT
  Severe aGHVD defined as grades 3-4. A stratified Cox regression analysis of time to CMV disease or PET following CMV reactivation prior to Day 180 post-HCT will be performed. The estimated hazard ratio and its 95% confidence interval will be calculated. Secondary analyses will include the Fine-Gray model for competing risk.
Incidence of severe adverse events (AEs) (safety in HCT-recipients) | Within 2 weeks from transplantation and up to 1 year post HCT
  Probably or definitely related to the vaccination per Common Terminology Criteria for Adverse Events version 5.0. A stratified Cox regression analysis of time to CMV disease or PET following CMV reactivation prior to Day 180 post-HCT will be performed. The estimated hazard ratio and its 95% confidence interval will be calculated. Secondary analyses will include the Fine-Gray model for competing risk.
Incidence of grade 3 and higher AEs (safety in HCT-donors) | Within 14 days
  A stratified Cox regression analysis of time to CMV disease or PET following CMV reactivation prior to Day 180 post-HCT will be performed. The estimated hazard ratio and its 95% confidence interval will be calculated. Secondary analyses will include the Fine-Gray model for competing risk.

SECONDARY OUTCOMES:
Time-to viremia (CMV-related events) | From transplantation to the date of two consecutive CMV quantitative polymerase chain reaction (qPCR) > 500 gc/mL/465 IU/mL or single event of CMV qPCR >1500 CMV gc/mL/1,395 IU/mL, assessed up to 1 year post HCT
  The number and percentage of recipients who receive treatment prior to the study recommended level of CMV viremia for PET will be tabulated by treatment group. Total days on antivirals for CMV reactivation (induction, maintenance, and total) will be assessed for each HCT recipient with treatment groups compared using Wilcoxson's rank sum test. Other characterizations of viremia and response to therapy will be descriptive in nature.
Duration of viremia (CMV-related events) | Up to 1 year post HCT
  The number and percentage of recipients who receive treatment prior to the study recommended level of CMV viremia for PET will be tabulated by treatment group. Total days on antivirals for CMV reactivation (induction, maintenance, and total) will be assessed for each HCT recipient with treatment groups compared using Wilcoxson's rank sum test. Other characterizations of viremia and response to therapy will be descriptive in nature.
Incidence of late CMV viremia (CMV-related events) | Between days 100-365 post HCT
  The number and percentage of recipients who receive treatment prior to the study recommended level of CMV viremia for PET will be tabulated by treatment group. Total days on antivirals for CMV reactivation (induction, maintenance, and total) will be assessed for each HCT recipient with treatment groups compared using Wilcoxson's rank sum test. Other characterizations of viremia and response to therapy will be descriptive in nature.
Use of antiviral drugs (CMV-related events) | Up to 1 year post HCT
  Triggered by clinically significant viremia or CMV disease.
Cumulative number of CMV specific antiviral treatment days (CMV-related events) | Up to 1 year post HCT
Incidence of CMV disease (CMV-related events) | Up to 1 year post HCT
Time to engraftment (transplant-related events) | Up to 1 year post HCT
Incidence of aGVHD and chronic GVHD (transplant-related events) | Up to 1 year post HCT
  Estimated using the Kaplan-Meier or Fine-Gray estimators, as appropriate, and compared using the log-rank test or the corresponding sub-distribution test of Gray.
Incidence of relapse (transplant-related events) | Up to 1 year post HCT
  Estimated using the Kaplan-Meier or Fine-Gray estimators, as appropriate, and compared using the log-rank test or the corresponding sub-distribution test of Gray.
Non-relapse mortality (transplant-related events) | Up to 1 year post HCT
All-cause mortality (transplant-related events) | Up to 1 year post HCT
Incidence of infections (transplant-related events) | Up to 1 year post HCT
  Estimated using the Kaplan-Meier or Fine-Gray estimators, as appropriate, and compared using the log-rank test or the corresponding sub-distribution test of Gray.
Levels and kinetics of CMV-specific T cell immunity, combined with immunophenotyping, and functional studies (immunological function) | Up to 1 year post HCT
  Generalized estimating equations will be used to estimate the effect of Triplex on log10-transformed concentration of CMV-specific T cells measured post-HCT. Initial regression model will include an indicator variable for Triplex vaccine status of the donor, study day as a categorical variable, and vaccine status by study day interaction term (saturated model). For each post-HCT day, difference in average log-10 concentration between study arms and its 95% confidence interval will be calculated. Primary analysis will include all post-HCT measurements. Additional analyses will be conducted in which measurements after CMV reactivation are excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Agrawal, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Northside Hospital, Atlanta, Georgia
  - DFCI/BWH Brigham and Women's Hospital, Boston, Massachusetts